CLINICAL TRIAL: NCT04194619
Title: A National Prospective Cohort for Pregnancies in Patients With Rare Vascular Anomalies: COGRare5 Study
Brief Title: Pregnancy in Women With Rare Multisystemic Vascular Diseases: COGRare5 Study
Acronym: COGRare5
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0380
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Vascular Anomaly; Osler Rendu Disease; Marfan Syndrome or Related; Lymphedema Primary; Arteriovenous Malformations; Cerebrospinal; Disorder
MeSH Terms: conditions — Vascular Malformations; Telangiectasia, Hereditary Hemorrhagic; Marfan Syndrome; Lymphedema; Arteriovenous Malformations; Central Nervous System Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Interview of women with a rare vascular disease through a phone questionnaire about severe and specific obstetrical complications during and after pregnancy.

SUMMARY:
There are no prospective studies of pregnancies for the diseases studied here in (Heredity Hemorrhagic Telangiectasia, Marfan syndrome or related, primary lower limb lymphedema, superficial arteriovenous malformations, and cerebro-spinal arteriovenous malformations) although complications of these can present life-threatening health problems for the mother and her baby.

The purpose of this National prospective study is to obtain greater insight into obstetrical complications associated with rare maternal vascular genetic disorders in order to improve prevention and to reduce risk of death.

In this context, experts and patient associations consider that there is a need to make real progress in the formulation of recommendations based on scientific data.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years and ≤45 years at the time of inclusion
* Pregnant and/or having given birth less than 1 month (≤ 30 days)
* Clinically and/or radiological and/or molecular biology diagnosis of a rare vascular disease before or during pregnancy or one month after delivery.
* Having been informed of all pertinent aspects of the study and provided oral non-opposition.

Exclusion Criteria:

* Any person not fulfilling the inclusion criteria or refusing to take part in the study.
* Major under legal protection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: This study describes severe and specific obstetrical complications during and after pregnancy (until 12 months postpartum) for the following pathologies: heredity hemorrhagic telangiectasia, marfan syndrome or related, primary lower limb lymphedema, superficial arteriovenous malformations or even cerebro-spinal arteriovenous malformations.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Occurrence of obstetrical complications among patients with rare vascular anomalies. | Every 3 months up to 21 months
  The primary outcome measure is the occurrence of specific and serious obstetrical complications during the pregnancy period and and after 12 months among patients with rare vascular anomalies, obtained via phone questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie DUPUIS-GIROD, MD, Principal Investigator — Service de Génétique - Hôpital Femme-Mère-Enfant - HCL
Locations (36):
- France (36):
  - Service de Médecine Interne et Maladies Vasculaires + Service Neuropédiatrie et neurochirurgie de l'enfant - CHU Angers, Angers
  - Service de Médecine interne et immunologie clinique + Service de Médecine Vasculaire - Hôpital Saint André, CHU de Bordeaux, Bordeaux
  - Service Pneumologie et Oncologie Thoracique - AP-HP Hôpital Ambroise Paré, Boulogne-Billancourt
  - Centre de Référence pour la maladie de Rendu-Osler - Service Génétique Clinique - Hôpital Femme-Mère-Enfant - Hospices Civils de Lyon, Bron
  - Service d'imagerie médicale - Neuroradiologie interventionnelle - Hôpital Neurologique P. Wertheimer - HCL, Bron
  - Service d'Imagerie Pédiatrique et Fœtale et Consultation Pluridisciplinaire des Angiomes - Hôpital Femme-Mère-Enfant - HCL, Bron
  - Service de Génétique, Hôpital Femme-Mère-Enfant, Bron
  - Service de Médecine Vasculaire - Hôpital de la Côte de Nacre, Caen
  - Service Médecine Interne Estaing CHU de Clermont-Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - CHU Dijon Bourgogne - Hôpital François Mitterrand, Dijon
  - Service de Médecine vasculaire et HTA - Hôpital Albert Calmette, CHRU de Lille, Lille
  - Service Médecine interne - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHU de Marseille - Hôpital de la Timone, Marseille
  - Service Médecine Interne - Hôpital Saint-Eloi, CHU de Montpellier, Montpellier
  - Service de neuroradiologie diagnostique et interventionnelle - CHU de Nancy, Hôpital St-Julien, Nancy
  - Service de Médecine Interne-Médecine Vasculaire, CHU de Nantes - Hôtel Dieu, Nantes
  - Unité de neuro-interventionnelle CHU Nice, Hôpital Pasteur 2, Nice
  - Service de dermatologie, CHU de Nice - Hôpital l'Archet 2, Nice
  - Service de Neuroradiologie - AP-HP - Paris (Hôpital Lariboisière), Paris
  - Service de Lymphologie - Hôpital Cognacq-Jay - Paris, Paris
  - Service de Cardiologie - Hôpital Bichat, AP-HP, Paris
  - Service de Neuroradiologie Interventionnelle - Fondation Adolphe de Rothschild, Paris
  - Service Radiologie-pneumologie interventionnelle - Hôpital Tenon AP-HP, Paris
  - Service de Génétique CHU de Poitiers, Poitiers
  - Service de Pneumologie CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Unité de Génétique médicale, CHU de Rennes, Hôpital Sud, Rennes
  - Service Médecine Interne - Médecine vasculaire - CHU de Rouen, Hôpital Charles Nicolle, Rouen
  - Service de Médecine Vasculaire et Thérapeutique, Explorations Fonctionnelles Vasculaires - CHU de Saint-Etienne - Hôpital Nord, Saint-Etienne
  - Clinique cardiologique et des maladies vasculaires CHU de Nantes, Hôpital G. R. LAENNEC, Saint-Herblain
  - Service Maladies vasculaires - HTA - NHC Pôle Médico-chirurgicale cardio-vasculaire, CHU de Strasbourg - Hôpital Civil, Strasbourg
  - CHU de Strasbourg, Hôpital de Hautepierre, Strasbourg
  - Service de Neuroradiologie Interventionnelle - Hôpital Foch, Suresnes
  - Service de Cardiologie _ Hôpital des Enfants (Purpan), Toulouse
  - Service de Médecine Interne + Service Médecine Vasculaire _ Hôpital RANGUEIL, Toulouse
  - Service Pneumologie, Hôpital Bretonneau, Centre Hospitalier Régional Universitaire de TOURS, Tours
  - CHU de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No